CLINICAL TRIAL: NCT05870254
Title: Exergaming With Immersive Virtual Reality to Improve Functional Abilities in People With Multiple Sclerosis
Brief Title: Exergaming With Immersive Virtual Reality For People With Multiple Sclerosis (ExeRVIEM)
Acronym: ExeRVIEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Collaborators: Asociación Viguesa de Esclerosis Múltiple de Pontevedra (Unknown)
Responsible Party: Principal Investigator, Pablo Campo-Prieto, Principal Investigator, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HEALTHYFIT-UVIGO 1/2023
Record Dates: First submitted 2023-03-22; First posted 2023-05-23 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis; Physical Therapy; Exercise; Virtual Reality Exposure Therapy; Rehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ExeRVIEM Protocol (Experimental): They will carry out the ExeRVIEM program for 8 weeks (2 times a week). Intervention based on exercise therapies with RVI software.
  Interventions: Other: ExeRVIEM Program; Other: Usual center program
- Usual Protocol (Active Comparator): They will carry out the usual protocol of Association
  Interventions: Other: Usual center program

INTERVENTIONS:
Other: ExeRVIEM Program — Virtual exercise based program
  Arms: ExeRVIEM Protocol
Other: Usual center program — Usual center cares

SUMMARY:
TITLE: Exergaming with Immersive Virtual Reality for people with Multiple Sclerosis

INTRO: Multiple Sclerosis (MS) is an autoimmune and chronic neurodegenerative pathology caused by loss of the myelin sheath in the nervous system, causing motor, cognitive, behavioral and sensory symptoms.

Conventional physiotherapy often includes exercise therapies, based on repetitive performances that can sometimes be unmotivating for patients. Immersive Virtual Reality could offer programs based on exercise (exergames) that are motivating, as well as appropriate to the therapeutic objectives of the target group. This tool has already been successfully tested in other groups (post stroke, Parkinson's,...) with promising results.

Our ExeRVIEM project (Exergaming with Immersive Virtual Reality in Multiple Sclerosis) represents a new strategy to improve functionality in people with MS, using an exercise program with Virtual Reality glasses.

HYPOTHESIS: The practice of the ExeRVIEM protocol based on physical function training in people with MS contributes to the maintenance and improvement of functional capacities, reducing the number of falls and increasing their personal autonomy.

GENERAL OBJECTIVES:

1.1 Design and implement an ExeRVIEM exercise program/protocol to improve balance in older people

1.2 Analyze the effects of this ExeRVIEM program/protocol, in the short and medium term in people who attend an Association of patients.

1.3 Identify if there is a relationship between the variables that induce frailty and functional dependence and the ExeRVIEM protocol.

SPECIFIC OBJECTIVES:

2.1 Determine and apply the ExeRVIEM protocol to explore differential effects for 6 minutes a day (2 days a week for 8 weeks).

2.1.1 Improving the functional independence and mobility of people by improving balance, reducing the risk of falls and the correct development of activities of daily living.

2.1.2 Gait improvement. 2.1.3 Improved functionality. 2.1.4 Improving grip strength. 2.1.5 Improving reaction times. 2.1.6 Improving the perception of fatigue

2.2 Determine the influence of parameters related to exposure to RVI.

2.2.1 Safety of the virtual reality exhibition 2.2.2 Usability of the virtual reality exhibition 2.2.3 Personal experiences and satisfaction of the virtual reality exhibition

METHODS:

Design: Randomized controlled trial. People diagnosed with MS who attend the AVEMPO VIGO center in Spain on a regular basis will be invited to participate in the study. After they meet the selection criteria, they will be assigned to an experimental group and a control group. Information on the sociodemographic characteristics and a clinical history of the participants will be collected.

Intervention: Two groups (experimental and control). The experimental group will carry out the ExeRVIEM protocol sessions (6 min) focused on the upper and lower limbs. (2 sessions per week for 8 weeks). All sessions will begin with a warm-up focused on stimulating coordination and joint mobilization, so that the body is predisposed both centrally and peripherally to carry out the session and will end with a stretching routine accompanied by breathing calm and controlled cycles. The session will be supervised by the center's physiotherapist or occupational therapist.

The control group will continue with the usual activities proposed by the center team.

Evaluations: 3 evaluations will be carried out: initial, final (at 8 weeks) and follow-up (one month after the end of the program).

The contents of the evaluations will be:

Patient characteristics: "Ad hoc" record sheet that will include data on age, sex, years since diagnosis, MS subtype, and drug treatment.

1. ExeRVIEM protocol. Safety (Simulator Sickness Questionnaire), Usability (System Usability Scale) and personal experiences (Game Experience Questionnaire and "ad hoc" interview notebook)
2. Balance, gait and risk of falling (Tinetti Test) 3. Functional mobility and lower limb strength (Five times sit to stand test) 4. Functional autonomy (Timed Up and Go Test- simple and cognitive) 5. Fatigue (Fatigue Severity Scale) 6 Handgrip (dynamometer) 7. Reaction time (Rezzil Software)

Hypothesis: Our findings aim to support the use of new health technologies in the field of rehabilitation and medical care for people with MS, achieving a feasible and safe Immersive Virtual Reality exergaming program.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with MS belonging to the AVEMPO VIGO Association
* Ages between 18-65 years
* Ability to stay on your feet and follow the intervention protocol and scheduled assessments

Exclusion Criteria:

* Medical report that advises against the practice of physical activity and exercise
* Uncontrolled outbreak of the disease
* Dizziness, vertigo or severe visual impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Balance, gait and risk of falling | pre-intervention
  TINETTI TEST
Balance, gait and risk of falling | immediately after the intervention
  TINETTI TEST
Balance, gait and risk of falling | 4 weeks after the intervention
  TINETTI TEST
functional autonomy | pre-intervention
  TIMED UP GO
functional autonomy | immediately after the intervention
  TIMED UP GO
functional autonomy | 4 weeks after the intervention
  TIMED UP GO
functional and cognitive autonomy | pre-intervention
  TIMED UP GO COGNITIVE
functional and cognitive autonomy | immediately after the intervention
  TIMED UP GO COGNITIVE
functional and cognitive autonomy | 4 weeks after the intervention
  TIMED UP GO COGNITIVE
functional mobility and lower limb strength | pre-intervention
  Five Times Sit to Stand Test
functional mobility and lower limb strength | immediately after the intervention
  Five Times Sit to Stand Test
functional mobility and lower limb strength | 4 weeks after the intervention
  Five Times Sit to Stand Test
Reaction Time | pre-intervention
  SOFTWARE REZZIL
Reaction Time | immediately after the intervention
  SOFTWARE REZZIL
Reaction Time | 4 weeks after the intervention
  SOFTWARE REZZIL
Fatigue | pre-intervention
  The Fatigue Severity Scale
Fatigue | immediately after the intervention
  The Fatigue Severity Scale
Fatigue | 4 weeks after the intervention
  The Fatigue Severity Scale

SECONDARY OUTCOMES:
Safety of the IVR intervention | immediately after the intervention
  Simulator Sickness Questionnaire
Usability of the IVR intervention | immediately after the intervention
  System Usability Scale
Satisfaction and experiences post IVR intervention | immediately after the intervention
  Game Experience Questionnaire-POST GAME MODULE

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - University of Vigo, Pontevedra, Galicia
  - University of Vigo, Pontevedra

IPD SHARING:
Plan to Share IPD: No